CLINICAL TRIAL: NCT05661435
Title: Utility of Remote Lung Auscultation in Transitions of Care After Pulmonary Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Utility of Remote Lung Auscultation in Transitions of Care After Pulmonary Exacerbations of COPD
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor Hold
Sponsor: Strados Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SL-RS-TJUH01
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Participants
  Interventions: Device: RESP Biosensor

INTERVENTIONS:
Device: RESP Biosensor — The RESP Biosensor will be placed on the patient for periodic recording of auscultory sound.
  Other Names: RESP

SUMMARY:
Listening to breath sounds with the stethoscope/auscultation is used by pulmonary physicians in conjunction with pulmonary function, signs and symptoms, oxygen saturation and diagnostic testing to admit, follow and discharge patients from hospital. Of these, only auscultation routinely ceases upon discharge from Hospital. Healthcare utilization statistics have shown that for more than a decade, readmission after discharge for an exacerbation of COPD or severe asthma (or chronic heart failure) remains a major problem. The Strados RESP Biosensor has been designed to extend the range of lung sound recording both geographically and temporally to improve the standard of care when access to continuous monitoring has been replaced by periodic or no monitoring. The primary purpose of this study is to assess the associations between RESP Biosensor-acquired lung findings and subjective measures of respiratory symptoms as measured by validated measurement tools, and objective measure of respiratory physiology as determined by home spirometry

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 35 and 75 with documented physician-diagnosed COPD
2. Hospitalization with a primary diagnosis of COPD with exacerbation or pneumonia.
3. Patient able and willing to provide informed consent.
4. Patient can follow study procedures, including instructions for self-placement and operation of device

   a. Patient has experience using a smartphone
5. Accessible by telehealth/telephone upon discharge
6. Patient is able and willing to return to study site for study follow-up visits as necessary

Exclusion Criteria:

1. Patient unable or unwilling to provide informed consent
2. Diagnosis of COPD is uncertain
3. Plan for discharge to location other than the patient's home (eg, Nursing Home, Rehabilitation facility)
4. Patient with end-stage medical condition with expected survival no more than 3 months
5. History of adverse reaction or allergy to TegaDerm®
6. Inaccessible by telehealth/telephone post discharge

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are admitted to the hospital for exacerbation of COPD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Statistically significant associations between RESP Biosensor-acquired lung findings and 1) subjective measure of respiratory symptoms measured by validated measurements tools and 2) home spirometry | Periodic recording over 24 hours for 30 days

SECONDARY OUTCOMES:
Univariate and multivariate assessment of predictors of 30 day respiratory-disease specific hospital readmission rate | Periodic recording over 24 hours for 30 days
Univariate and multivariate assessment of predictors of 30 day total respiratory exacerbation rate (moderate + severe) | Periodic recording over 24 hours for 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided